CLINICAL TRIAL: NCT06563648
Title: The Effect of Local Cold Application and ShotBlocker Use in Subcutaneous Injection on Injection Pain and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bornova No. 25 Mevlana Family Health Center (Other)
Collaborators: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Ince, research assistant faculty of nursing principles, Ege University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Ege
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pain; Satisfaction, Patient
Keywords: Subcutaneous injection; shotblocker; cold application; low molecular weight heparin; pain; satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ShotBlocker group (Experimental): A ShotBlocker was placed on the arm of the patients in the ShotBlocker group during the injection, and the injection was performed from the part where the opening was located by lightly pressing with the fingertips throughout the injection.
  Interventions: Other: shotblocker
- ShotBlocker placebo group (Experimental): During the injection, the back side of the ShotBlocker was placed on the arm of the patients in the ShotBlocker placebo group and the injection was performed by gently pressing with the fingertips throughout the injection.
  Interventions: Other: ShotBlocker placebo group
- Local cold application group (Experimental): Local cold application was applied to the arm of the patients in the local cold application group for five minutes using a cold pack,and then the injection was performed.
  Interventions: Other: local cold application
- control group (No Intervention): Patients in the control group were injected with a routine subcutaneous injection procedure.

INTERVENTIONS:
Other: shotblocker — A ShotBlocker was placed on the arm of the patients in the ShotBlocker group during the injection, and the injection was performed from the part where the opening was located by lightly pressing with the fingertips throughout the injection.
  Arms: ShotBlocker group
Other: local cold application — Local cold application was applied to the arm of the patients in the local cold application group for five minutes using a cold pack, and then the injection was performed.
  Arms: Local cold application group
Other: ShotBlocker placebo group — During the injection, the back side of the ShotBlocker was placed on the arm of the patients in the ShotBlocker placebo group and the injection was performed by gently pressing with the fingertips throughout the injection.
  Arms: ShotBlocker placebo group

SUMMARY:
The research was conducted as a single-blind, randomized controlled, experimental study to determine the effect of ShotBlocker and local cold application on pain and patient satisfaction in subcutaneous heparin injection.

DETAILED DESCRIPTION:
The research was conducted as a single-blind, randomized controlled, experimental study to determine the effect of ShotBlocker and local cold application on pain and patient satisfaction in subcutaneous heparin injection. The research was conducted with 208 patients hospitalized in the Cardiology and Internal Medicine clinics at Izmir Atatürk Training and Research Hospital between April 2022 and April 2024. Patients were assigned to four groups: ShotBlocker (n=52), ShotBlocker placebo (n=52), local cold application (n=52) and control (n=52) groups using the randomization algorithm.

A ShotBlocker was placed on the arm of the patients in the ShotBlocker group during the injection, and the injection was performed from the part where the opening was located by lightly pressing with the fingertips throughout the injection. During the injection, the back side of the ShotBlocker was placed on the arm of the patients in the ShotBlocker placebo group and the injection was performed by gently pressing with the fingertips throughout the injection. Local cold application was applied to the arm of the patients in the local cold application group for five minutes using a cold pack, and then the injection was performed. Patients in the control group were injected with a routine subcutaneous injection procedure. In all groups, the injection took 30 seconds and was performed by researcher. At the first minute after the injection, the patients were evaluated about the pain they felt during the injection and their satisfaction with the injection by a different reseacher. Data were collected by face-to-face interview technique using an informed consent form, individual identification form, visual analog scale and visual patient satisfaction scale. Ethics committee permission, institutional permission and written permission from the patients were obtained for the implementation of the research. Number, percentage, median, mean, and standard deviation, Mann Whitney U test, Kolmogorov-Smirnov test, Kruskal Wallis H test, Bonferroni and chi-square test were used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Enoxaparin sodium 1x1 0.6 ml. SC treatment
* Over 18 years of age
* No vision or hearing problems
* No scar tissue, incision, lipodystrophy or infection at the injection site

Exclusion Criteria:

* Underwent mastectomy
* Not being voluntering

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | At the first minute after the injection, the patients were evaluated about the pain they felt during the injection by a different reseacher.
  The VAS is used to assess the severity of acute pain. It is mostly a horizontal or vertical line 100 mm long, starting with "no pain" and ending with "unbearable pain". It is used to convert some values that cannot be measured numerically to a numerically usable form

SECONDARY OUTCOMES:
Visual patient satisfaction scale | At the first minute after the injection, the patients were evaluated their satisfaction with the injection by a different reseacher.
  The visual patient satisfaction scale combines the characteristics of the well-known VAS. At one end of the scale is the phrase "I am not satisfied at all", and at the other end is the phrase "I am very satisfied". It is mostly a horizontal or vertical line 100 mm long.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university nursing faculty, Izmir, Bornova, Turkey (Türkiye)

REFERENCES:
- [Background] Usach I, Martinez R, Festini T, Peris JE. Subcutaneous Injection of Drugs: Literature Review of Factors Influencing Pain Sensation at the Injection Site. Adv Ther. 2019 Nov;36(11):2986-2996. doi: 10.1007/s12325-019-01101-6. Epub 2019 Oct 5. PMID 31587143
- [Background] Wang H, Guan J, Zhang X, Wang X, Ji T, Hou D, Wang G, Sun J. Effect of Cold Application on Pain and Bruising in Patients With Subcutaneous Injection of Low-Molecular-Weight Heparin: A Meta-Analysis. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620905349. doi: 10.1177/1076029620905349. PMID 32372652
- [Background] Woodley WD, Morel DR, Sutter DE, Pettis RJ, Bolick NG. Clinical evaluation of large volume subcutaneous injection tissue effects, pain, and acceptability in healthy adults. Clin Transl Sci. 2022 Jan;15(1):92-104. doi: 10.1111/cts.13109. Epub 2021 Nov 10. PMID 34268888